CLINICAL TRIAL: NCT04046861
Title: "Influence of High Vitamin C Dose on Lactate During Extracorporeal Circulation for Heart Surgery and During the 24 Hours Thereafter." (double Blind Prospective Randomised Study)
Brief Title: Influence of High Vitamin C Dose on Lactate During and After Extracorporeal Circulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Centre Maribor (Other)
Responsible Party: Principal Investigator, Andreja Möller Petrun, MD, PhD, MD, PhD, Assistant professor, University Medical Centre Maribor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: UKC-MB-KME-20/19
Record Dates: First submitted 2019-07-27; First posted 2019-08-06 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Hyperlactatemia; Cardiac Disease; Bypass Complication; Valve Disease, Heart; Vitamin C
Keywords: cardiac surgery; cardiopulmonary bypass; hyperlactatemia; vitamin C
MeSH Terms: conditions — Hyperlactatemia; Heart Diseases; Heart Valve Diseases | interventions — Ascorbic Acid; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vitamin C (Active Comparator): 2g vitamin C (ascorbic acid) iv before cardiopulmonary bypass, 2 g vitamin C iv before removing the aortic clamp, 1g vitamin C iv 8 h after aortic clamp removal and every 8 h thereafter(2 times)
  Interventions: Dietary Supplement: ascorbic acid,
- Placebo (saline) (Placebo Comparator): placebo (saline) iv before cardiopulmonary bypass, placebo before removing the aortic clamp, placebo iv 8 h after aortic clamp removal and every 8 h (2 times)
  Interventions: Other: Placebo (saline)

INTERVENTIONS:
Dietary Supplement: ascorbic acid, — The vitamin C group will get high dose of intravenous vitamin C (ascorbic acid) before starting cardiopulmonary bypass, before removing aortic clamp and every 8 hours thereafter for additionaly 24 hours
  Other Names: Vitamin C
  Arms: Vitamin C
Other: Placebo (saline) — The placebo group will get saline before starting cardiopulmonary bypass, before removing aortic clamp and every 8 hours thereafter for additionaly 24 hours
  Arms: Placebo (saline)

SUMMARY:
The aim of our study is to find out whether high doses of vitamin C before cardiopulmonary bypass and during the first 24 hours after that have and impact of lowering the incidence of hyperlactatemia.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years old patients with cardiac disease needing surgery (coronary bypass, valve replacement)

Exclusion Criteria:

* dementia
* kidney stones
* dialysis
* haemochromatosis
* thalassemias
* G-6-P deficiency

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Concentration of lactate | up to 30 hours
  Measuring the concentration of lactate before cardiopulmonary bypass, after aortic clamp removal, at ICU admission,then every 6 hours

SECONDARY OUTCOMES:
dose of noradrenaline and other vasopressors | up to 36 hours
  The need for noradrenaline and other vasopressors (e.g. vasopresin) during the surgery and in the 24-hours after the end of the surgery

OTHER OUTCOMES:
Concentration of glucose | up to 30 hours
  Measuring the concentration of glucose before cardiopulmonary bypass, after aortic clamp removal, at ICU admission, then every 6 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Department od anesthesiology, intensive care and pain management, Maribor, Slovenia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Laffey JG, Boylan JF, Cheng DC. The systemic inflammatory response to cardiac surgery: implications for the anesthesiologist. Anesthesiology. 2002 Jul;97(1):215-52. doi: 10.1097/00000542-200207000-00030. No abstract available. PMID 12131125
- [Background] Bronicki RA, Hall M. Cardiopulmonary Bypass-Induced Inflammatory Response: Pathophysiology and Treatment. Pediatr Crit Care Med. 2016 Aug;17(8 Suppl 1):S272-8. doi: 10.1097/PCC.0000000000000759. PMID 27490610
- [Background] Hall R. Identification of inflammatory mediators and their modulation by strategies for the management of the systemic inflammatory response during cardiac surgery. J Cardiothorac Vasc Anesth. 2013 Oct;27(5):983-1033. doi: 10.1053/j.jvca.2012.09.013. Epub 2012 Dec 29. No abstract available. PMID 23276596
- [Background] Roy J, Galano JM, Durand T, Le Guennec JY, Lee JC. Physiological role of reactive oxygen species as promoters of natural defenses. FASEB J. 2017 Sep;31(9):3729-3745. doi: 10.1096/fj.201700170R. Epub 2017 Jun 7. PMID 28592639
- [Background] Koekkoek WA, van Zanten AR. Antioxidant Vitamins and Trace Elements in Critical Illness. Nutr Clin Pract. 2016 Aug;31(4):457-74. doi: 10.1177/0884533616653832. Epub 2016 Jun 16. PMID 27312081
- [Background] Stoppe C, McDonald B, Benstoem C, Elke G, Meybohm P, Whitlock R, Fremes S, Fowler R, Lamarche Y, Jiang X, Day AG, Heyland DK. Evaluation of Persistent Organ Dysfunction Plus Death As a Novel Composite Outcome in Cardiac Surgical Patients. J Cardiothorac Vasc Anesth. 2016 Jan;30(1):30-8. doi: 10.1053/j.jvca.2015.07.035. Epub 2015 Jul 29. PMID 26847748
- [Background] Ellenberger C, Sologashvili T, Cikirikcioglu M, Verdon G, Diaper J, Cassina T, Licker M. Risk factors of postcardiotomy ventricular dysfunction in moderate-to-high risk patients undergoing open-heart surgery. Ann Card Anaesth. 2017 Jul-Sep;20(3):287-296. doi: 10.4103/aca.ACA_60_17. PMID 28701592
- [Background] Lomivorotov VV, Efremov SM, Kirov MY, Fominskiy EV, Karaskov AM. Low-Cardiac-Output Syndrome After Cardiac Surgery. J Cardiothorac Vasc Anesth. 2017 Feb;31(1):291-308. doi: 10.1053/j.jvca.2016.05.029. Epub 2016 Jul 29. No abstract available. PMID 27671216
- [Background] Hill A, Wendt S, Benstoem C, Neubauer C, Meybohm P, Langlois P, Adhikari NK, Heyland DK, Stoppe C. Vitamin C to Improve Organ Dysfunction in Cardiac Surgery Patients-Review and Pragmatic Approach. Nutrients. 2018 Jul 27;10(8):974. doi: 10.3390/nu10080974. PMID 30060468
- [Background] O'Connor E, Fraser JF. The interpretation of perioperative lactate abnormalities in patients undergoing cardiac surgery. Anaesth Intensive Care. 2012 Jul;40(4):598-603. doi: 10.1177/0310057X1204000404. PMID 22813486
- [Background] Gladden LB. Lactate metabolism: a new paradigm for the third millennium. J Physiol. 2004 Jul 1;558(Pt 1):5-30. doi: 10.1113/jphysiol.2003.058701. Epub 2004 May 6. PMID 15131240
- [Background] Chatham JC. Lactate -- the forgotten fuel! J Physiol. 2002 Jul 15;542(Pt 2):333. doi: 10.1113/jphysiol.2002.020974. No abstract available. PMID 12122132
- [Background] Levy B. Lactate and shock state: the metabolic view. Curr Opin Crit Care. 2006 Aug;12(4):315-21. doi: 10.1097/01.ccx.0000235208.77450.15. PMID 16810041
- [Background] Levy B, Perez P, Perny J, Thivilier C, Gerard A. Comparison of norepinephrine-dobutamine to epinephrine for hemodynamics, lactate metabolism, and organ function variables in cardiogenic shock. A prospective, randomized pilot study. Crit Care Med. 2011 Mar;39(3):450-5. doi: 10.1097/CCM.0b013e3181ffe0eb. PMID 21037469
- [Background] Maillet JM, Le Besnerais P, Cantoni M, Nataf P, Ruffenach A, Lessana A, Brodaty D. Frequency, risk factors, and outcome of hyperlactatemia after cardiac surgery. Chest. 2003 May;123(5):1361-6. doi: 10.1378/chest.123.5.1361. PMID 12740248
- [Background] Levy B, Sadoune LO, Gelot AM, Bollaert PE, Nabet P, Larcan A. Evolution of lactate/pyruvate and arterial ketone body ratios in the early course of catecholamine-treated septic shock. Crit Care Med. 2000 Jan;28(1):114-9. doi: 10.1097/00003246-200001000-00019. PMID 10667509
- [Background] Frei B, Stocker R, England L, Ames BN. Ascorbate: the most effective antioxidant in human blood plasma. Adv Exp Med Biol. 1990;264:155-63. doi: 10.1007/978-1-4684-5730-8_24. PMID 2244489
- [Background] Berger MM, Oudemans-van Straaten HM. Vitamin C supplementation in the critically ill patient. Curr Opin Clin Nutr Metab Care. 2015 Mar;18(2):193-201. doi: 10.1097/MCO.0000000000000148. PMID 25635594
- [Background] Tyml K. Vitamin C and Microvascular Dysfunction in Systemic Inflammation. Antioxidants (Basel). 2017 Jun 29;6(3):49. doi: 10.3390/antiox6030049. PMID 28661424
- [Background] Oudemans-van Straaten HM, Spoelstra-de Man AM, de Waard MC. Vitamin C revisited. Crit Care. 2014 Aug 6;18(4):460. doi: 10.1186/s13054-014-0460-x. PMID 25185110
- [Background] Dingchao H, Zhiduan Q, Liye H, Xiaodong F. The protective effects of high-dose ascorbic acid on myocardium against reperfusion injury during and after cardiopulmonary bypass. Thorac Cardiovasc Surg. 1994 Oct;42(5):276-8. doi: 10.1055/s-2007-1016504. PMID 7863489